CLINICAL TRIAL: NCT01001442
Title: A Phase I/IIa Multi-Dose Escalation Study to Evaluate Maximum Tolerated Dose (MTD), Pharmacokinetics (PK), Safety and Efficacy of BT062 in Subjects With Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Safety and Dose Determining Multi-dose Study of BT062 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotest Pharmaceuticals Corporation (Industry)
Collaborators: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 975
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Relapsed; Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — indatuximab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BT062 (Experimental): BT062 was to be administered as single-dose IV infusions via a 0.22 μm in-line filter preferably in a forearm vein, according to medically accepted procedures on Days 1, 8, and 15 of each 28-day cycle. Alternatively BT062 may have been administered through a central venous line or a peripherally inserted central catheter (PICC). Other administration routes were only to be allowed after approval from Biotest. Each subject was to be monitored carefully for the effects of exposure to BT062. No subject was to have received more than 3 doses of BT062 per 28-day treatment cycle.
  Interventions: Drug: BT062

INTERVENTIONS:
Drug: BT062 — intravenous administration
  Other Names: Indatuximab ravtansine

SUMMARY:
This Phase I/IIa clinical study is to test safety and anti-tumor activity of BT062 to define the best dose in treating patients with relapsed or refractory multiple myeloma with multiple doses of BT062.

DETAILED DESCRIPTION:
Phase I/IIa, open-label, 3 + 3 multi-dose escalation study. The Phase I part of the study was to include the dose escalation cohort; a conventional dose escalation design, following 3 + 3 rules was chosen to define the MTD.

The Phase IIa part was to include the MTD/recommended phase II dose (RPTD) expansion cohort in which descriptive statistical methods for evaluation of response, time to event endpoints, and safety were to be performed.

35 subjects in the Safety population, 34 subjects in the ITT and PP populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active multiple myeloma according to the International Myeloma Working Group diagnostic criteria
* Relapsed or relapsed/refractory multiple myeloma
* Previous treatment with both an immunomodulator and a proteosome inhibitor therapy
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (Zubrod) ≤ 2
* Ability to understand and willingness to sign a written informed consent document
* Ability to adhere with the study visit schedule and other protocol procedures
* Life expectancy of ≥ 12 weeks
* Normal organ and marrow function

Exclusion Criteria:

* Chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to day 1 or those who have not recovered from AEs due to agents administered more than 3 weeks earlier
* Treatment with another investigational agent during the study or within 4 weeks before day 1
* Major surgery within 4 weeks before day 1 (this does not include placement of vascular access device or tumor biopsies)
* Antineoplastic therapy with biological agents within 2 weeks before day 1
* Known HAHAs, HACAs, or HAMAs in response to previous MAb therapy
* Previous treatment with BT062
* Malignancy within 3 years before day 1, other than the trial indication multiple myeloma and excluding treated non-melanoma skin cancer, superficial bladder cancer and carcinoma in-situ of the cervix
* Severe diseases of skin, colon, esophagus, or eye within 1 year before day 1, as judged by the Investigator
* Severe infections necessitating use of antibiotics / antivirals during the screening period
* Clinically relevant active infection including active hepatitis B or C or human immunodeficiency virus (HBV, HCV, or HIV) or any other concurrent disease which, in the judgment of the investigator, would make the subject inappropriate for enrollment into this study
* Acute or relevant abnormalities in electrocardiogram (ECG), as judged by the Investigator. These abnormalities can be defined as recent myocardial infarction, uncontrolled cardiac arrhythmias and/or pronounced disturbances of the electrical conduction system of the heart.
* Significant cardiac disease such as recent myocardial infarction (≤ 6 months prior to day 1), unstable angina, uncontrolled congestive heart failure, uncontrolled hypertension (recurrent or persistent increases in systolic blood pressure ≥ 180 mm Hg or diastolic blood pressure ≥ 110 mm Hg), uncontrolled cardiac arrhythmias, grade 3 (Lown Criteria) or greater cardiac toxicity from prior chemotherapy
* History of clinically significant drug or alcohol abuse
* Unwillingness or inability to adhere to the requirements of the study
* Concomitant therapy with corticosteroids (except as indicated in low dose for other medical conditions such as inhaled steroid for asthma, topical use, or as premedication for administration of certain medications (including BT062) or blood products and for treatment of infusion reactions if needed)
* Concomitant antineoplastic therapies including chemotherapy, radiotherapy, or biological agents during the study
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he or she are included in the study
* Breast-feeding
* Unwillingness to use an effective contraceptive method during the study and at least 3 months after administration of study drug - unless subject is naturally infertile. (Acceptable contraceptive methods include oral or injectable contraceptives, intrauterine devices (IUD), double-barrier method, contraceptive patch, surgical sterilization, or condoms).
* Positive serum or urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C. Anderson, MD, Study Director — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Mount Sinai School of Medicine, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Intention-to-treat (ITT) population included all subjects who were enrolled in the study and received at least 1 dose of BT062 and who had any post-Baseline evaluations or data. One subject did not have at least one post-injection assessment of the treatment response and was excluded from both the ITT and PP populations (n = 34).
Groups:
- BT062 40 mg/m²: 40 mg/m² BT062 was administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
- BT062 50 mg/m²: 50 mg/m² BT062 was administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
- BT062 65 mg/m²: 65 mg/m² BT062 was administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
- BT062 80 mg/m²: 80 mg/m² BT062 was administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
- BT062 100 mg/m²: 100 mg/m² BT062 was administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
- BT062 120 mg/m²: 120 mg/m² BT062 was administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
- BT062 140 mg/m²: 140 mg/m² BT062 was administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
- BT062 160 mg/m²: 160 mg/m² BT062 was administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
Period: Overall Study
Arm/Group | BT062 40 mg/m² | BT062 50 mg/m² | BT062 65 mg/m² | BT062 80 mg/m² | BT062 100 mg/m² | BT062 120 mg/m² | BT062 140 mg/m² | BT062 160 mg/m²
Started | 4 | 3 | 4 | 3 | 4 | 3 | 10 | 4
Completed | 4 | 3 | 4 | 3 | 2 | 3 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Population: ITT: The Intention-to-treat (ITT) population included all subjects who were enrolled in the study and received at least 1 dose of BT062 and who had any post-Baseline evaluations or data. One subject did not have at least one post-injection assessment of the treatment response and was excluded from both the ITT and PP populations (n = 34).
Groups:
- Total: Total of all reporting groups
Arm/Group | BT062 40 mg/m² | BT062 50 mg/m² | BT062 65 mg/m² | BT062 80 mg/m² | BT062 100 mg/m² | BT062 120 mg/m² | BT062 140 mg/m² | BT062 160 mg/m² | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 10 | 4 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 2 | 2 | 1 | 3 | 2 | 3 | 17
  >=65 years | 3 | 0 | 2 | 1 | 2 | 0 | 8 | 1 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (15.56) | 55.3 (7.64) | 64.3 (9.39) | 60.7 (4.51) | 64.3 (8.02) | 55.3 (5.03) | 66.8 (8.80) | 61.5 (9.98) | 63.5 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 2 | 1 | 5 | 2 | 18
  Male | 2 | 0 | 2 | 2 | 1 | 2 | 5 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 3 | 3 | 3 | 3 | 3 | 9 | 3 | 31
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 1 | 7
  White | 4 | 3 | 3 | 3 | 2 | 2 | 6 | 3 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 3 | 3 | 3 | 10 | 4 | 34

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLT) - Number of Participants With at Least 1 DLT
Description: The primary safety variable was to determine the incidence of DLTs in subjects with relapsed or relapsed/refractory multiple myeloma treated with BT062.
Time Frame: Starting with first study drug administration until 30-day follow-up visit (average 4.99 months)
Population: The Safety population included all subjects who were enrolled and received at least
  1 dose of BT062 (n = 35).
Measure: Count of Participants; unit: Participants
Groups:
- Total: BT062 administration (all dose levels)
Arm/Group | BT062 40 mg/m² | BT062 50 mg/m² | BT062 65 mg/m² | BT062 80 mg/m² | BT062 100 mg/m² | BT062 120 mg/m² | BT062 140 mg/m² | BT062 160 mg/m² | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 4 | 3 | 10 | 4 | 35
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 5

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The Phase I part of the study was to include the dose escalation cohort; a conventional dose escalation design, following 3 + 3 rules was chosen to define the MTD.
  Only DLTs occurring in cycle 1 for each subject were counted in the dose escalation decisions.
  Three subjects were treated at the first or newest dose level as available. If none of the 3 subjects experienced a DLT during Cycle 1, three subjects could be treated at the next dose level as available.
  In case of a DLT the cohort was expanded to up to 6 subjects. If not more than 1 of these 6 subjects experienced a DLT during Cycle 1, a first subject could be treated at the next dose level.
  If 2 or more of the 6 subjects experienced a DLT during Cycle 1 the dose escalation was stopped.
  The highest dose level at which < 2 of 6 subjects experienced a DLT is defined as the MTD.
Time Frame: First 28-day cycle
Measure: Number; unit: mg/m²
Arm/Group | BT062
Number analyzed (Participants) | 35
mg/m² | 140

3. Secondary Outcome: Qualitative and Quantitative Toxicities of BT062
Description: Qualitative and quantitative toxicities assessed by incidence of adverse events and by clinically significant changes in the patient's physical examination, vital signs, and clinical laboratory results.
  The incidence of treatment emergent adverse events (TEAEs), including serious adverse events (SAEs).
Time Frame: Starting with first study drug administration until 30-day follow-up visit (average 4.99 months)
Population: Safety Population: The Safety population included all subjects who were enrolled and received at least 1 dose of BT062 (n = 35).
Measure: Count of Participants; unit: Participants
Arm/Group | BT062 40 mg/m² | BT062 50 mg/m² | BT062 65 mg/m² | BT062 80 mg/m² | BT062 100 mg/m² | BT062 120 mg/m² | BT062 140 mg/m² | BT062 160 mg/m² | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 4 | 3 | 10 | 4 | 35
Participants
  At least one SAE | 2 | 0 | 0 | 2 | 2 | 1 | 5 | 2 | 14
  At least one treatment related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3

4. Secondary Outcome: Multi-dose Pharmacokinetics Properties of BT062 - Cmax
Description: Multi-dose Pharmacokinetics properties of BT062 after intravenous (IV) Administration of escalating doses of BT062 as assessed by measuring intact BT062 conjugate.
  Please note that not all subjects reached Cycle 4 due to early termination . A lower number of samples could be analyzed for Cycle 4.
Time Frame: Starting with first study drug administration until 30-day follow-up visit (average 4.99 months).
Population: as for outcome 3
Measure: Median (Full Range); unit: ng/ml
Arm/Group | BT062 40 mg/m² | BT062 50 mg/m² | BT062 65 mg/m² | BT062 80 mg/m² | BT062 100 mg/m² | BT062 120 mg/m² | BT062 140 mg/m² | BT062 160 mg/m²
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 4 | 3 | 10 | 4
ng/ml
  BT062 plasma concentration Cycle 1 - Cmax: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 9 | 2
  BT062 plasma concentration Cycle 1 - Cmax | 13409.0 [3725 to 15888] | 10156.0 [7108 to 14028] | 26229.0 [17114 to 58194] | 21498.0 [18827 to 31112] | 51593.0 [36526 to 93993] | 61190.0 [29640 to 66623] | 48463.0 [32175 to 70734] | 62876.5 [47149 to 78604]
  BT062 plasma concentration Cycle 4 - Cmax: number analyzed (Participants) | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  BT062 plasma concentration Cycle 4 - Cmax | 9427.0 [9427 to 9427] | 14193.0 [14193 to 14193] | 27770.5 [23740 to 31801] | 38144.0 [38144 to 38144] | 92046.0 [92046 to 92046] | 96178.0 [42123 to 150233] | 50073.0 [50073 to 50073] | 79248.0 [79248 to 79248]

5. Secondary Outcome: Anti-tumor Activity of BT062 in Subjects With Relapsed or Relapsed/Refractory Multiple Myeloma by Number of Participants With Objective Response(ORR) and/or Clinial Benefit(CBR) Based on the International Myeloma Working Group Uniform Response Criteria
Description: sCR:CR+normal FLC+absence of clonal cells in BM; CR:Negative immunofixation,disappearance of soft tissue plasmacytomas +≤5% plasma cells in BM+normal FLC; VGPR:M-protein detectable by immunofixation,not on electrophoresis or 90% or greater reduction in serum M-protein+urine M-protein level <100mg per 24h,>90% decrease in the difference between involved/uninvolved FLC; PR:≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200 mg per 24 h or ≥50% decrease in the difference between involved/uninvolved FLC or ≥50% reduction in plasma cells, provided baseline bone marrow plasma cell percentage was ≥30%, ≥50% size reduction of soft tissue plasmacytomas; MR:25%-49% reduction of serum M-protein+reduction in 24h urinary M-protein by 50-89%(still >200 mg/24h),25-49% soft tissue plasmacytomas size reduction,no increase in size or number of lytic bone lesions; SD:no response or PD ORR: %of subjects with MR+PR+VGPR+CR+sCR CBR:ORR + %of subjects with SD.
Time Frame: On day 1 of each treatment cycle (on a monthly basis) starting with first study drug administration until Close Out visit (average 3.84 months).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BT062 40 mg/m² | BT062 50 mg/m² | BT062 65 mg/m² | BT062 80 mg/m² | BT062 100 mg/m² | BT062 120 mg/m² | BT062 140 mg/m² | BT062 160 mg/m² | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 10 | 4 | 34
Participants
  Objective Response rate: yes | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Objective Response rate: no | 4 | 3 | 4 | 2 | 3 | 3 | 9 | 4 | 32
  Clinical Benefit rate: yes | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 5
  Clinical Benefit rate: no | 4 | 3 | 4 | 2 | 3 | 2 | 9 | 2 | 29

6. Secondary Outcome: Time to Progression (TTP), Progression Free Survival (PFS) and Overall Survival (OS)
Description: Progressive disease
  Requires any one or more of the following:
  Increase of ≥ 25% from baseline in
  * Serum M-component and/or (the absolute increase must be ≥ 0.5 g/dL) (increases of ≥ 1 g/dL are sufficient to define relapse if starting M-component is ≥ 5 g/dL).
  * Urine M-component and/or (the absolute increase must be ≥ 200mg/24h).
  Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL.
  Bone marrow plasma cell percentage: the absolute % must be ≥ 10% (relapse form CR as a 5% cutoff instead of 10%).
  Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas.
  Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/l) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: Starting with first study drug administration until death or 3 years from first study treatment.
Population: The Intention-to-treat (ITT) population included all subjects who were enrolled in the study and received at least 1 dose of BT062 and who had any post-Baseline evaluations or data (n = 34).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BT062
Number analyzed (Participants) | 34
months
  TTP | 3 [1.1 to 4.4]
  PFS | 3 [1.1 to 3.9]
  OS | 26.7 [13.2 to 42.4]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were to be documented during the entire study period including the 30 day follow up (average 4.99 months).
Arm/Group | BT062 40 mg/m² | BT062 50 mg/m² | BT062 65 mg/m² | BT062 80 mg/m² | BT062 100 mg/m² | BT062 120 mg/m² | BT062 140 mg/m² | BT062 160 mg/m² | Total
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/3 | 1/4 | 1/3 | 1/10 | 1/4 | 4/35
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 0/4 | 2/3 | 2/4 | 1/3 | 5/10 | 2/4 | 14/35
Other Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 3/4 | 2/3 | 3/4 | 3/3 | 8/10 | 3/4 | 28/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT062 40 mg/m² (N=4) | BT062 50 mg/m² (N=3) | BT062 65 mg/m² (N=4) | BT062 80 mg/m² (N=3) | BT062 100 mg/m² (N=4) | BT062 120 mg/m² (N=3) | BT062 140 mg/m² (N=10) | BT062 160 mg/m² (N=4) | Total (N=35)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EXTRAOCULAR MUSCLE PARESIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRAIN MASS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
ALVEOLITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PALMAR-PLANTAR / ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT062 40 mg/m² (N=4) | BT062 50 mg/m² (N=3) | BT062 65 mg/m² (N=4) | BT062 80 mg/m² (N=3) | BT062 100 mg/m² (N=4) | BT062 120 mg/m² (N=3) | BT062 140 mg/m² (N=10) | BT062 160 mg/m² (N=4) | Total (N=35)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 1 (2) | 3 (4) | 1 (1) | 11 (14)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 3 (4)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 4 (5)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 4 (5)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 2 (7) | 3 (3) | 3 (4) | 13 (21)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 8 (9)
FATIGUE (General disorders) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (5) | 2 (2) | 1 (2) | 12 (17)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
INFUSION SITE ERYTHEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 7 (7)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
INFUSION RELATED (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 3 (4) | 1 (2) | 6 (10)
AMYLASE INCREASED (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (5)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 9 (11)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
BLOOD URIC ACID INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
OCCULT BLOOD POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 6 (11)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 2 (2) | 7 (11)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
DYSURIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 5 (7)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 3 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 5 (7)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Part of CTA:The Investigator or any Site employee, consultant or admitting physician to the Site or Study Team member is not allowed to make any publication of any Study Data, information, results, or similar information without the review and comment of SPONSOR. As the Study is part of a multi-center trial, and the Investigator/site agree that no publication by Site/Investigator of the results of the Study conducted at the Site shall be made before the first multi-centre publication.